CLINICAL TRIAL: NCT07109583
Title: Effects of Dinner Timing on Eating Behaviour, Physical Activity and Metabolic Health
Brief Title: Impact of Dinner Timing on Human Behaviours and Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202203HM008-2
Record Dates: First submitted 2025-06-26; First posted 2025-08-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Delayed Dinner Intervention
Keywords: Eating behaviour; Physical activity; Metabolic health
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early dinner (Experimental): Consume dinner between 17:30 and 19:00 for one week
  Interventions: Behavioral: Early dinner
- Delayed dinner (Experimental): Consume dinner between 20:30 and 22:00 for one week
  Interventions: Behavioral: Delayed dinner

INTERVENTIONS:
Behavioral: Early dinner — Consume dinner between 17:30 and 19:00 for a week
  Arms: Early dinner
Behavioral: Delayed dinner — Consume dinner between 20:30 and 22:00 for a week
  Arms: Delayed dinner

SUMMARY:
The aim of this project is to investigate the impact of dinner timing on eating behaviors, physical activity and metabolic healthy in healthy adults

DETAILED DESCRIPTION:
In the early dinner trial, participants will be required to eat dinner between 17:30 and 19:00 for a week. In the delayed dinner trial, participants will be required to eat dinner between 20:30 and 22:00 for a week. During the intervention, energy intake (3 days of weekday and 1 day of weekend), physical activity (7 days), glucose concentrations (7 days) and sleep (7 days) will be monitored continuously for both early and delayed dinner.

After intervention, body composition, cognition, food preference, metabolic health and resting metabolic rate will be measured.

ELIGIBILITY:
Inclusion Criteria:

* No regular exerciser in the last 3 months.
* BMI between 18.5-27 kg/m².
* Regular habit of eating three meals per day, with dinner consumed between 17:00 and 20:00.
* No intentional weight change (>3%) in the past 3 months.
* No special dietary practices (e.g., intermittent fasting).
* Regular sleep (22:00-01:00), at least 6.5 hours per night.
* Non-smoker and non-alcoholic.
* Willing to maintain stable lifestyle and comply with protocol.

Exclusion Criteria:

* Pregnancy, preparing for pregnancy or menopause.
* Personal history of/existing diabetes, cardiovascular disease or metabolic diseases.
* Diagnosed sleep disorders.
* Taking medications influencing glucose metabolism.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Glucose responses | During 7 days of early dinner and 7 days of delayed dinner intervention
  Changes in blood glucose responses between early and delayed dinner intervention
Eating behaviour | During early dinner and delayed dinner intervention (3 days of weekday and 1 day of weekend)
  Meal choice (i.e., energy intake in kcal) between early and delayed dinner intervention

SECONDARY OUTCOMES:
Sleep duration | During 7 days of early dinner and 7 days of delayed dinner intervention
  Changes in sleep duration between early and delayed dinner intervention using MotionWatch
Sleep quality | During 7 days of early dinner and 7 days of delayed dinner intervention
  Changes in sleep quality (efficiency, %) between early and delayed dinner intervention using MotionWatch
Physical activity level | During 7 days of early dinner and 7 days of delayed dinner intervention
  Changes in physical activity level (minutes) between early and delayed dinner intervention
Physical activity intensity | During 7 days of early dinner and 7 days of delayed dinner intervention
  Changes in physical activity intensity (%) between early and delayed dinner intervention using wearable product
Cognitive performance | Before and after early and delayed dinner intervention
  Changes in computerized cognitive performance (accuracy in %) after early and delayed dinner intervention
Food preference tests | Before and after early and delayed dinner intervention
  Changes in food preference after early and delayed dinner intervention
Resting resting metabolic rate | Before and after early and delayed dinner intervention
  Changes in resting metabolic rate (kcal) after early and delayed dinner intervention
Body composition | Before and after early and delayed dinner intervention
  Changes in body composition (fat mass in kg and percentage) after early and delayed dinner intervention using InBody
Blood pressure | Before and after early and delayed dinner intervention
  Changes in blood pressure (diastolic and systolic blood pressure in mmHg) after early and delayed dinner intervention
Pulse wave velocity | Before and after early and delayed dinner intervention
  Changes in pulse wave velocity (meter per second) after early and delayed dinner intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chen, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan